CLINICAL TRIAL: NCT00747786
Title: An Observational, Multicentre, Open Label, Non Interventional Programme to Assess the Long-Term Safety and Efficacy of Somatuline Autogel in the Treatment of Neuroendocrine Tumours When Administered by Patients or Their Partners ("Home Injection Group") or Administered by Healthcare Professionals
Brief Title: Non Interventional Post Marketing Programme in Neuroendocrine Tumours
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: Y-97-52030-215
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study, is to assess the safety and local tolerability of the long-term use of Somatuline Autogel when administered by patients or their partners ("Home Injection Group") and the safety and local tolerability in patients receiving their injection from a healthcare professional (HCP) ("Reference Group").

ELIGIBILITY:
Inclusion Criteria:

* The patient must give written (personally signed and dated) informed consent for their data to be included in the database for this Post Marketing Surveillance programme and any subsequent analysis.
* The patient must have been receiving treatment with Somatuline Autogel at a stable dose for at least 4 months.
* The patient must have a diagnosis of neuroendocrine tumours
* The patient must be at least 18 years of age
* For patients receiving or intending to receive Somatuline Autogel by home injection:

  * The patient must be able to store Somatuline Autogel safely in a refrigerator in their own home and either collect it from their GP/Pharmacy on a monthly basis, or receive the medication by a home delivery service.

Exclusion Criteria:

* The patient is pregnant or breast-feeding, unless continued treatment with Somatuline Autogel is clearly needed (as determined by the treating clinician).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neuroendocrine tumours seen in routine clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-12; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
safety and local tolerability of Somatuline Autogel when administered by patients or their partners or from a healthcare professional | End of observational period

SECONDARY OUTCOMES:
efficacy of Somatuline Autogel | End of observational period
training requirements for patients / partners to perform home injection of Somatuline Autogel | End of observational period
acceptability of home injections to patients, partners and healthcare professionals | End of observational period

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (5):
- United Kingdom (5):
  - University Hospital of Wales, Cardiff
  - Aintree University Hospital, Liverpool
  - Royal Free Hospital, London
  - St. Bartholomew's Hospital, London
  - Royal Hallamshire Hospital, Sheffield